CLINICAL TRIAL: NCT00003154
Title: Phase II Trial of 9-Aminocamptothecin (9-AC) Colloidal Dispersion (CD) 120-Hour Continuous Intravenous Infusion in Advanced Non-Small Cell Lung Cancer
Brief Title: Chemotherapy in Treating Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Nathan Levitan, MD, Ireland Cancer Center At University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU1597; U01CA063200 (NIH); P30CA043703 (NIH); CWRU-1597 (Other: Case Comprehensive Cancer Center); NCI-T97-0024
Record Dates: First submitted 1999-11-01; First posted 2004-05-19 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: aminocamptothecin colloidal dispersion — 120 hour continuous infusion of aminocamptothecin colloidal dispersion (AC/CD) once a week for 2 weeks, followed by 1 week of rest. Patients are assessed after every 2 courses of therapy. Treatment with aminocamptothecin continues indefinitely if there is tumor shrinkage or stable disease and no significant toxicity is experienced. Patients are followed every 3 months.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of aminocamptothecin in treating patients with stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether aminocamptothecin colloidal dispersion (AC/CD) administered as a 120 hour weekly infusion is an effective treatment for advanced non-small cell lung cancer. II. Observe any toxicities associated with this treatment in this patient population.

OUTLINE: Patients receive a 120 hour continuous infusion of aminocamptothecin colloidal dispersion (AC/CD) once a week for 2 weeks, followed by 1 week of rest. Patients are assessed after every 2 courses of therapy. Treatment with aminocamptothecin continues indefinitely if there is tumor shrinkage or stable disease and no significant toxicity is experienced. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 19-36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed measurable stage IIIB or IV non-small cell lung cancer No brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: WBC at least 3500/mm3 Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT and SGPT no greater than 2.5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 2.5 times ULN Renal: Creatinine no greater than 1.5 mg/dL Creatinine clearance at least 60 mL/min Calcium and electrolytes normal Other: No other malignancy within past 5 years except curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix Not pregnant or nursing No active infections or other serious medical conditions

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 2 weeks since prior radiotherapy No prior radiotherapy to site(s) of measurable disease Surgery: At least 3 weeks since any prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 1998-01; Primary Completion 2001-04 (Actual); Study Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
Study the effectiveness of aminocamptothecin in treating patients with stage III or stage IV non-small cell lung cancer. | 120 hour continuous infusion once a week for 2 weeks, followed by 1 week of rest. Patients are assessed after every 2 courses of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Levitan, MD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States